CLINICAL TRIAL: NCT04157049
Title: Alpha-1 Research Registry Protocol
Brief Title: Alpha-1 Research Registry
Status: Recruiting | Type: Observational
Sponsor: Alpha-1 Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Alpha-1 Registry Protocol
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: AATD; ALPHA 1; COPD; AAT; ZZ; MZ; CARRIER; MM; MS; PiZZ
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alpha-1 Diagnosed Individuals: Larger patient cohorts are needed to support the clinical trials coming in the next 3-5 years. Despite widespread invitations to the Alpha-1 community from the Alpha-1 Foundation Research Registry, it is estimated that the Alpha-1 Foundation Research Registry now contains <40% of the identified PiZZ individuals in the US.
- Carriers of Alpha-1: Larger patient cohorts are needed to support the clinical trials coming in the next 3-5 years. Despite widespread invitations to the Alpha-1 community from the Alpha-1 Foundation Research Registry, it is estimated that the Alpha-1 Foundation Research Registry now contains <40% of the identified PiZZ individuals in the US.

SUMMARY:
The Alpha-1 Research Registry is a confidential database made up of individuals diagnosed with Alpha-1 Antitrypsin Deficiency (Alpha-1) and individuals identified as Alpha-1 carriers. The Registry was established to facilitate research initiatives and promote the development of improved treatments and a cure for Alpha-1.

DETAILED DESCRIPTION:
The purpose and goal of the Alpha-1 Research Registry (Registry, or group of patients) will be to obtain uniform, longitudinal (over the course of time), complete and accurate data that can be organized, and made available for the public to query. The collective number of Registry members enables investigators to enroll sufficient subjects to carry out their studies. The community benefits from having more research and potential therapies performed in their disease. Regular updates from patients will give objective data-points to measure the progression of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Alpha-1 Antitrypsin Deficiency (PiZZ, PiZNull, PiSZ etc.)
* Alpha-1 carriers (PiMZ, PiMS etc.)

Exclusion Criteria:

* Failure to provide informed consent
* Normal healthy individuals (MM)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The current protocol seeks to enroll 4,000 individuals of all age, race, and sex.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2029-06-20 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
Establish the Alpha-1 Research Registry using REDCap | 2 years
  To gather accurate patient data for longitudinal prospective follow up/analysis of Alpha-1 progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Alpha-1 Foundation, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided